CLINICAL TRIAL: NCT00654667
Title: Mechanisms of Metabolic Regulation of Resveratrol on Humans With Metabolic Syndrome.
Acronym: RSV
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participant enrollment
Sponsor: University of California, San Francisco (Other)
Responsible Party: Marlene Berro, UCSF
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTSI - SOS
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Insulin Resistance
Keywords: Resveratrol; Insulin Resistance; Metabolic Syndrome; Sirtuin 1; IGF-1; Satiety; Leptin; Adiponectin
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Experimental 1 (Experimental): Resveratrol
  Interventions: Drug: Resveratrol

INTERVENTIONS:
Drug: Placebo — Placebo, no active drug, take 5 capsules by mouth daily for one month
  Arms: 2
Drug: Resveratrol
  Arms: Experimental 1

SUMMARY:
Sirtuin activators may prove useful in treating age-related diseases and extending lifespan in humans. Resveratrol (RSV), a polyphenol found in red wine, has been shown in vitro to enhance SIRT1 activity. RSV is associated with some of the beneficial effects of red wine or the "French Paradox". Recently RSV has been associated with increasing lifespan in mice on a high calorie diet and improved metabolic profile and activity levels. The effect of this small molecule in humans is unknown. Preclinical observations suggest that RSV is safe and has enormous potential in the treatment of obesity and insulin resistance in humans. This pilot study will examine the effect of RSV on improving the metabolic profile of adults with insulin resistance. Specifically, this randomized double blind placebo controlled study will examine the effects of 4 weeks of supplementation with RSV 5.0 grams daily, compared to placebo control (PC) on the metabolic profile of 36 men and women over the age of 50 with insulin resistance (IR) consuming a typical western diet consisting of at least 40% calories from fat.

DETAILED DESCRIPTION:
Hypotheses for this study:

4 weeks of supplementation with RSV 5.0 grams daily compared to placebo control in individuals with insulin resistance will: 1) Increase insulin sensitivity (assessed by the insulin sensitivity index as derived from glucose and insulin levels obtained during a 2 hour oral glucose tolerance test (OGTT)and insulin growth factor (IGF)-1 levels) 2) Improve cholesterol metabolism (lower LDL, raise HDL and lower triglyceride (TG) levels); and 3) physical activity levels measured by pedometer and 7 day physical activity recall (PAR).

Secondary hypotheses are: Treatment with RSV 5.0 grams daily in individuals with IR will result in: 1)No change in energy intake as measured by food intake by 3 day food diary; 2)No change in body fat mass or distribution (via dual x-ray absorptiometry (DEXA), body mass index (BMI) and waist-to-hip ratio; and 3)Improved Quality of life as assessed by SF-36, compared to PC group.

We will also examine self-reported appetite and satiety as well as biomarkers leptin and adiponectin in the RSV versus PC group. Finally, we will examine the effects of RSV on hepatic (serum Ala aminotransferase, asp aminotransferase, lactate dehydrogenase, alkaline phosphatase, bilirubin, albumin), pancreatic (serum amylase) and renal (BUN and creatinine), function and red blood cell count (CBC with differential) in the IR compared to the PC group.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 50 years or older
2. Women ages 50 years and older who are postmenopausal, defined as no menses for the previous 12 months
3. BMI 25 to 35
4. Waist-to-hip circumference ratios for men >0.95, for women >0.85
5. HOMA-IR score from fasting plasma glucose and serum insulin levels >2.7
6. A diet consisting of > 40% calories from fat; and
7. Sedentary, defined as no formal exercise program and less than 30 minutes physical activity weekly.

Exclusion Criteria:

1. Active malignancy or tumor or other condition that would severely limit life expectancy
2. Any type of major surgery during the last 3 months
3. Psychiatric disorders with currently active manifestations
4. Insulin-dependent diabetes
5. Any chronic medications except for hormone replacement therapy. Vitamin supplements (of any type) are not allowed during the study, but are acceptable if the participant agrees to a 2 week washout period before participation in the study
6. Active symptoms suggestive of an acute coronary syndrome or decompensated heart failure
7. Currently on low fat diet or special diet (i.e. weight loss)
8. Excessive alcohol intake (>3 glasses of wine/1 six pack of beer daily)
9. Concurrent participation in any drug studies or studies that require sample of a body fluid (or having finished in the past 6 months)
10. Non-English speakers
11. Abnormal LFTs.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity (assessed by the insulin sensitivity index as derived from glucose and insulin levels obtained during a 2 hour oral glucose tolerance test (OGTT)1, 2 and insulin growth factor (IGF)-1 levels3 | one month

SECONDARY OUTCOMES:
Improve cholesterol metabolism (lower LDL, raise HDL and lower triglyceride (TG) levels); and 3) physical activity levels measured by pedometer and 7 day physical activity recall (PAR) | one month

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, California, United States